CLINICAL TRIAL: NCT03617133
Title: Image Guided Intensity Modulated External Beam Radiochemotherapy and MRI Based Adaptive BRAchytherapy in Locally Advanced CErvical Cancer
Brief Title: Image Guided IMRT, Radiochemotherapy and MRI-based IGABT in Locally Advanced Cervical Cancer
Acronym: EMBRACEII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other); Odense University Hospital (Other); North Estonia Medical Centre (Other); Institut Bergonié (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); University Hospital Heidelberg (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Oslo University Hospital (Other); Institute of Oncology Ljubljana (Other); Complejo Hospitalario de Navarra (Other); Hospital Clinic of Barcelona (Other); Skane University Hospital (Other); Region Örebro County (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Radiotherapiegroep (Other); Leiden University Medical Center (Other); Maastro Clinic, The Netherlands (Other); UMC Utrecht (Other); The Netherlands Cancer Institute (Other); Radboud University Medical Center (Other); Catharina Ziekenhuis Eindhoven (Other); Erasmus Medical Center (Other); Cambridge University Hospitals NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); The Christie NHS Foundation Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Royal Marsden NHS Foundation Trust (Other); Cross Cancer Institute (Other); McGill University (Other); Princess Margaret Hospital, Canada (Other); Tom Baker Cancer Centre (Other); Loyola University Chicago (Other); M.D. Anderson Cancer Center (Other); University of Pittsburgh (Other); Pamela Youde Nethersole Eastern Hospital (Other); Tuen Mun Hospital (Other Government); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Tata Memorial Centre (Other); Chulalongkorn University (Other); Siriraj Hospital (Other); Liverpool Hospital, Sydney (Unknown); Maisonneuve-Rosemont Hospital (Other); National Cancer Institute, Slovakia (Other Government); Institut Català d'Oncologia (Other); Ludwig-Maximilians - University of Munich (Other); Mount Vernon Cancer Centre (Unknown); St Thomas' Hospital, London (Other)
Responsible Party: Principal Investigator, Richard Pötter, Principal investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMBRACE 2
Record Dates: First submitted 2018-07-13; First posted 2018-08-06 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Interventional, observational, validation study to EMBRACE I
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard arm (Other): General and specific aims of EMBRACEII as well as the multiple quantitative hypotheses are based on technical data, dose volume parameters and clinical results of the prospective observational study EMBRACEI (NCT00920920, 3 year data 2015) and the retrospective RetroEMBRACE (3/5 year data 2015). The performance of EMBRACE II interventions and clinical outcome in terms of disease- (local, nodal, systemic control, OS, CSS) and morbidity-outcome (various organs and endpoints) is thus based on recent clinical evidence with radiochemotherapy and image guided adaptive brachytherapy. The expected effect of EMBRACE II interventions on clinical outcome is estimated from comparative analyses of interventions in subgroups of Retro-/EMBRACE (partly published). Based on the Retro-/EMBRACE benchmark, the estimated outcome including a confidence interval is quantified for each clinical endpoint in the overall cohort as well as different subgroups for an overall expected patient number of 1000.
  Interventions: Radiation: Increased use of IC/IS technique in BT; Radiation: Reduction of vaginal source loading; Radiation: Systematic utilisation of IMRT; Radiation: Utilisation of daily IGRT (set-up according to bony structures); Radiation: EBRT target concept related to the primary tumor (CTV-T) and internal motion; concepts for OAR contouring; Radiation: EBRT dose prescription and reporting; Radiation: Adaptation of EBRT nodal elective CTV according to risk of nodal and systemic recurrence; Drug: Systemic application of simultaneous chemotherapy; Other: Reduction of overall treatment time

INTERVENTIONS:
Radiation: Increased use of IC/IS technique in BT — In EMBRACE II, the improved therapeutic window (through increased application of IC/IS) will be exploited for tumour dose-(de-)escalation and/or OAR dose de-escalation. In tumours with large residual CTVHR volumes at time of brachytherapy, dose-escalation has the potential to improve local control significantly. In limited size CTVHR volumes dose-de-escalation will be performed since dose de-escalation has minor impact on local control while it has potential to reduce morbidity. The strategy of EMBRACEII is to aim for an application of the IC/IS technique in at least 20% of the patients in each institution. The threshold of 20% is relevant for a classical stage distribution of ~20% IB, ~50% IIB, ~20% IIIB and ~10% others. If a given patient population includes significantly higher proportions of limited or extensive disease, the threshold of 20% IC/IS applications must be adapted.
Radiation: Reduction of vaginal source loading — A multicenter investigation in 50 EMBRACE patients from 3 institutions (Mohamed SM. et al, in submission 2015) shows that reduced loading in ring/ovoids and increased loading in tandem (and needles when available) can be applied without compromising CTVHR and GTVres dose. Decrease of relative vaginal loading from a mean of 50% to 33% had potential to reduce ICRU recto-vaginal dose by a mean of 4±4Gy, and furthermore, bladder and rectum doses could be reduced by 2-3Gy with the same re-arrangement of loading. Similar evidence is available from a study on simulation of different intracavitary standard loading patterns in EMBRACE patients, where it was shown that limited size tumours could often be covered by tandem loading alone (Nkiwane KS. et al. 2013).
Radiation: Systematic utilisation of IMRT — Many institutions deliver 3D conformal radiotherapy (3D CRT) based on a four-field box technique although IMRT has been available for a number of years. The practice in EMBRACEI has been utilisation of IMRT and 3D CRT in 27% and 73% of the patients, respectively. However, EMBRACE morbidity data as well as data published by Mundt et al (Mundt AJ. et al. 2003) indicate that IMRT significantly reduces the incidence of bowel morbidity, and therefore IMRT is considered as instrumental for reducing the incidence of bowel morbidity and with a potential also to be beneficial for urinary morbidity.
Radiation: Utilisation of daily IGRT (set-up according to bony structures) — PTV margins of 10 mm to the elective lymph node target are currently applied in many institutions. This margin is related to set-up uncertainties with patient positioning performed based on skin marks. However, currently, most institutions have in-room imaging available which makes it possible to perform daily imaging and couch correction according to fusion on bony anatomy. With daily imaging, bony image fusion, and couch correction, a margin reduction from 10mm to 5mm can be performed without compromising target coverage (Laursen LV. et al. 2012). The 5mm margin reduction has potential to decrease the volume irradiated to 43Gy by approximately 500cm, which is expected to decrease bowel morbidity by ~50%.
Radiation: EBRT target concept related to the primary tumor (CTV-T) and internal motion; concepts for OAR contouring — New target concepts are introduced for EBRT related to primary tumor: initial CTV-T, initial CTV-HR, initial CTV-LR and ITV-LR. Use of this novel contouring approach in conjunction with available MRI allows to target safely the visible tumor (CTV-T) and the high risk region (CTV-HRintitial) while consenting for dose to a low risk region (CTV-LRinitial). Anatomical changes due to organ filling variation and cervix/uterus position are considered. ITV-LR is outlined using planning scan and MR images in patients with MRI in treating position while a fixed margin is added to the CTV-LR initial in patients with only diagnostic MRI. New concepts are introduced for OAR contouring. Bowel loops are outlined in one volume restricted to the outer contour, including the mesenterium, for better approximation of the bowel volume and dose constraints. Rectum/sigmoid structures are contoured distinctly. Vaginal lower border is 2,5cm from the caudal extend of the tumor (2cm ITV-LR initial + 0,5cm PTV).
Radiation: EBRT dose prescription and reporting — There is currently a significant variation with regard to EBRT dose and fractionation in the EMBRACE study with doses ranging from 45Gy to 50Gy and being delivered in 25-30 fractions. Furthermore, there is a wide variety of lymph node boosting strategies. In EMBRACEII, the EBRT dose and fractionation to the elective lymph node CTV and initial CTV-T is fixed at 45Gy in 25 fractions, and lymph node boosting must be performed as a simultaneous integrated boost. The dose de-escalation from 50Gy to 45Gy has potential to reduce morbidity. A system of reporting dose to targets and OARs is introduced in terms of dose volume parameters and a system of point dose reporting for the vagina.
Radiation: Adaptation of EBRT nodal elective CTV according to risk of nodal and systemic recurrence — EMBRACEII applies a risk adapted target concept for nodal CTV. This target concept is based on pattern of nodal recurrence analysis which shows 50% of recurrences beyond the classical L5/S1 cranial pelvic field border. A target volume "Large Pelvis" is defined for intermediate risk patients and includes internal, external, common iliac, obturator and presacral nodes. For high risk patients, defined as common iliac or >2 nodes involved, the para-aortic region is included. For low risk patients, defined as stage IA/IB1/IIA1, N0, small cell carcinoma (SCC), no uterine invasion, "Small Pelvis" is defined which is "Large Pelvis" without common iliac nodes. Intermediate risk is defined as not high and not low risk.
Drug: Systemic application of simultaneous chemotherapy — According to international standard and evidence, simultaneous chemotherapy (CHT) (min. 5x40 mg/m2 cis Platinum) was prescribed in the EMBRACE protocol for all patients, who qualify for its administration. Certain rules were given for adaption according to international guidelines. 90-95% of EMBRACE patients received simultaneous CHT. Most of the EMBRACE cohort is consecutive patients representing the cervix cancer patient population in the respective centers. About 70% of patients received ≥5 cycles, while 30% received 0-4 cycles. CHT has impact on systemic control, which is pronounced in high risk patients (node positive and/or stage III/IV) with a 20% difference in systemic recurrence. A center effect has been found in the ability to administer chemotherapy with 15-85% of the patients receiving ≥5 cycles of CHT. To reach optimal outcome, particularly in the high risk group, the EMBRACEII protocol also focusses on appropriate administration of CHT following international guidelines.
Other: Reduction of overall treatment time — Several studies indicate that maintaining an overall treatment time (OTT) of <=50 days is important for local control. RetroEMBRACE data confirms that OTT remains of importance in the realm of IGABT. As there is significant variation of OTT across patients and institutions in retroEMBRACE, the EMBRACEII study aims to reduce the OTT so that the majority of patients (>80%) will adhere to the <=50 day threshold. The measures to reduce OTT in EMBRACE is to systematically apply 25 fractions of EBRT including lymph node boost, and furthermore to carefully plan the BT schedule, so that brachytherapy is delivered towards the end of EBRT and/or directly after EBRT.

SUMMARY:
The research group on adaptive image-guided radiotherapy for locally advanced cervical carcinoma completed the protocol for the EMBRACE II study in October 2018. This study will be carried out in the next few years at the University Clinic for Radiotherapy at the Medical University of Vienna and other international partner institutes. EMBRACE II builds on the findings of the current EMBRACE study. These are already implemented in everyday clinical practice in order to further improve the accuracy of the entire therapy of cervical carcinomas, using state-of-the-art techniques of tele- and brachytherapy. The aim of the EMBRACE II study is to maintain and enhance the excellent local tumor control as well as the nodal and systemic control for all tumor stages while minimizing the adverse reaction rates for all affected organs (rectum, sigmoid, urinary bladder, and vagina) to increase the quality of life of patients with cervical carcinomas.

DETAILED DESCRIPTION:
The standard treatment of locally advanced cervical cancer is radio-chemotherapy including external beam radiotherapy (EBRT), brachytherapy (BT) and concomitant chemotherapy with weekly Cisplatin. Image Guided Adaptive Brachytherapy (IGABT), with repetitive MRI regarded as gold standard, is increasingly recognized as the new paradigm replacing 2D BT and spreading throughout the world. This spread is at present predominantly in Europe, North America and in many places in Asia. The Gyn GEC ESTRO Recommendations I-IV have been used as the conceptual frame for these developments during the last decade and are now embedded into the new ICRU/GEC ESTRO report 88 (International Commission on Radiation and Units) which is being published in 2015.

Beside increasing mono-institutional clinical experience - also reported in literature - there is increasing clinical evidence and analyses from multi-institutional studies, in particular RetroEMBRACE (n=731) and EMBRACE (n>1350) about dose volume effects and outcome. The mature RetroEMBRACE clinical outcome data and dose volume effect analysis for disease outcome show an improved excellent local and pelvic control and survival and significant dose volume effects for IGABT. Overall treatment time was found to have significant impact on local control, and in addition, volume effects of EBRT were found (IMRT vs. 3D CRT) with impact on morbidity and quality of life. Furthermore, dose effects of chemotherapy (≥5 cycles) were found to have impact on survival in advanced disease. Comprehensive analyses from both large patient cohorts reveal further relevant treatment parameters with major impact on disease outcome, morbidity and quality of life. In the international community the results from the EMBRACE studies are regarded as benchmark for future clinical research in this field. Based on the large success of the RetroEMBRACE and EMBRACE studies, the EMBRACE study and research group decided to continue the clinical research work and to initiate a consecutive EMBRACE II study with interventions derived from the evidence collected within the EMBRACE studies.

INTERVENTIONS, AIMS AND HYPOTHESES

The EMBRACE II interventions address local, nodal and systemic treatment as well as exposure of organs at risk:

* Increased use of IC/IS (intracavitary/interstitial) technique in BT
* Reduction of vaginal source loading
* Systematic utilisation of IMRT
* Utilisation of daily IGRT (set-up according to bony structures)
* EBRT target concept related to the primary tumour; concepts for organ at risk (OAR) contouring
* EBRT dose prescription and reporting
* Adaptation of EBRT nodal elective CTV according to risk of nodal and systemic recurrence
* Systematic application of simultaneous chemotherapy
* Reduction of overall treatment time

The general aims of the EMBRACE II study are:

* To systematically apply IMRT with daily IGRT as well as advanced image guided adaptive BT in a prospective multi-centre setting
* To systematically implement a dose prescription protocol for IGABT
* To implement systematic contouring, prescription and reporting for EBRT CTV and OARs.
* To administer EBRT in different targets which are adapted to the risk of nodal and systemic failure: to improve para-aortic and
* systemic control in high risk patients and not to decrease lymph node control in low risk and intermediate risk patients
* To systematically administer simultaneous chemotherapy to EBRT to reach prescribed dose in as many patients as possible, in particular in high risk patients
* To benchmark an outstanding high level of local, nodal and systemic control as well as survival with application of advanced EBRT, BT and chemotherapy within limited overall treatment time
* To benchmark a low incidence of intermediate and major morbidity as well as a high level of quality of life with application of advanced EBRT, BT and chemotherapy

Beside these general aims, there is a significant number of specific aims which refer to the prospective validation of dose volume parameters from the EMBRACE analyses (e.g. dose escalation for large tumors with increased application of IC/IS techniques), to explore and evaluate dose volume parameters for EBRT and to identify prognostic parameters.

General and specific hypotheses were formulated for the various interventions (BT, EBRT, chemotherapy) and endpoints (disease, morbidity, quality of life).

TYPE OF DESIGN The study is a multicenter prospective interventional study with some areas for observational research (e.g. dose-volume histogram (DVH) for IMRT). Reporting on the key patient, tumor, treatment and outcome parameters is mandatory including disease, morbidity and quality of life. Sub-studies as on adaptive IMRT and translational research are optional for cooperation between individual departments. Patient registration and reporting will be performed by the individual investigator via the internet to a central database.

PATIENTS TO BE INCLUDED Patients with newly biopsy proven squamous carcinoma, adenocarcinoma or adeno-squamous carcinoma of the uterine cervix, International Federation of Gynecology and Obstetrics (FIGO) stage IB, IIA, IIB, IIIA, IIIB and IVA (and nodal status according to TNM) in whom definitive radio-chemotherapy with curative intent is planned are qualified for the study. Treatment has to include IGABT with MRI and IMRT with IGRT and ≥5 cycles of cis-Platin. Patients with para-aortic metastatic nodes (stage IVB) to the level of L2 are also eligible but patients with further dissemination are not (M0). Patient work up and staging includes as a minimum patient characteristics with performance status and blood tests (e.g. haemoglobin, lymphocytes), tumor status (biopsy), gynaecological examination, MRI of the pelvis, abdominal CT or MRI, whole body FDG PET-CT (preferably) or at least chest CT. Further investigations are applied if necessary (e.g. cystoscopy, rectoscopy) or done according to institutional practice (e.g. laparoscopic lymph node assessment). Baseline morbidity scoring and quality of life questionnaire are mandatory.

TREATMENT OF PATIENTS IN THE TRIAL All patients will receive both EBRT and concomitant chemotherapy and BT. Summation of EBRT and BT doses will be performed by calculation of a biologically equivalent dose in 2 Gy per fraction (EQD2) using the linear-quadratic model with alpha/beta = 10 Gy for tumour effects and alpha/beta = 3 Gy for late normal tissue damage. The repair half time is assumed to be 1.5 hrs. EBRT has to be delivered as IMRT/VMAT (Volumetric Modulated Arc Therapy) with daily cone beam CT (IGRT) in 25 fractions with 1.8 Gy to a total dose of 45 Gy given in 5 weeks. Target definition is MRI based (initial GTV) for the CTV-T with an initial HR and LR CTV-T and an ITV-T (Internal Target Volume). CT or MRI based nodal Target (CTV-E) is according to risk of nodal spread "Small Pelvis", "Large Pelvis" or "Large Pelvis + Para-aortic Region". Overall CTV/ITV to PTV margin is 5 mm. Involved nodes are boosted preferably based on Positron Emission Tomography (PET) CT with 10-15 Gy and treated as simultaneous integrated boost within 5 weeks (2.2-2.4 Gy per fraction). A range for DVH parameters for the various OARs - contoured according to specific protocols - is taken into account for treatment planning. The LR CTV-T and the CTV- E will be treated with 45 Gy by use of EBRT (PTV45). Maximal treatment time including both EBRT and BT is 50 days. Brachytherapy is prescribed with dose escalation for advanced disease with large adaptive CTV-THR including IC/IS techniques and dose de-escalation for limited size CTV-THR to spare organs at risk and in particular the upper vagina. The primary imaging method is MRI with the applicator in place which enables definition of the relevant volumes of interest directly on the images for treatment planning: GTVres, adaptive CTVHR, CTVIR and organ volumes. The applicator and the reference points are reconstructed in the same image series. All treatment plans have to be optimized to achieve defined planning aims for dose and volume parameters for tumor (D98 for GTVres) and target volumes (e.g. D90-95 Gy for adaptive CTV-THR) and for 2cm3 reference volumes for OARs (e.g. <80 Gy for bladder, <65 Gy for rectum) and for vaginal reference points (recto-vaginal point < 65 Gy, PIBS). If the planning aims cannot be achieved, limits for the finally prescribed dose levels are defined for GTVres, CTVHR, CTVIR, point A, bladder, rectum, sigmoid bowel and vagina. Planning aim doses and limits for the finally prescribed dose levels are based on the experience of the previous retroEMBRACE and EMBRACE trials. For chemotherapy weekly concomitant Cisplatin (40 mg/m2) for 5-6 courses is standard unless chemotherapy is precluded by patient age, co-morbidity and toxicity. Aim is to apply minimum 5 cycles of cis-Platin, in particular in advanced disease.

QUALITY ASSURANCE Only approved departments and investigators can enroll patients into the protocol. This approval is under the responsibility of the study coordinators. The approved departments are at present those that have contributed continuously to EMBRACE in a considerable number of patients. These departments have to go additionally through a QA procedure for IMRT/IGRT. New departments will have to go through a quality assurance (QA) procedure both for IGABT and IMRT/IGRT. Approval requires a compliance questionnaire, successful training, registration and submission of cases and positive evaluation by the study coordinators for each centre. There is no formal on site monitoring, but patient files and treatment plans must be kept at least until closure of the protocol and final analysis of the results is obtained. Continuous data monitoring is performed through the study offices in Vienna and Aarhus and through Utrecht for the centres in the Netherlands. Continuous education will be offered through ACT and annual workshops and EMBRACE meetings.

OUTCOME MEASURES Local and nodal (pelvic) control within the specific EBRT and BT targets (HR-CTV-T, IR-CTV, LR CTV-T; CTV-E, CTV-N) and morbidity related to OAR in the pelvis and the para-artic region as well as overall survival, cancer specific survival and systemic control are the primary outcome measures. All endpoints will be evaluated by actuarial statistics. Morbidity will be scored by use of the Common Terminology Criteria for Adverse Events (CTCAE v3.0/4.0). QoL will also be systematically recorded in all patients.

EVALUATION OF OUTCOME MEASURES Tumor and nodal remission status (complete, uncertain complete, partial, stable & progressive disease) will be evaluated 3 months after treatment by pelvic (para-aortic, CT) MRI and gynaecological examination. Regular follow-up including gynaecological examination will then be instituted with planned appointments 6, 9, 12, 18, 24, 30, 36, 48 and 60 months after treatment. Pelvic (para-aortic, CT) MRI will be repeated at 12 months after treatment or in case of suspected recurrence. Morbidity and quality of life will be scored systematically at base line and at each time point during follow-up.

SAMPLE SIZE AND DATA MATURITY The study aims at recruiting 1000 patients in 4 years and to follow them for at least 5 years to allow for a meaningful assessment of the endpoints by univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the uterine cervix considered suitable for curative treatment with definitive radio-(chemo)therapy including MRI guided BT
* Positive biopsy showing squamous-cell carcinoma, adenocarcinoma or adeno-squamous cell carcinoma of the uterine cervix.
* Staging according to FIGO and TNM guidelines
* MRI of pelvis at diagnosis is performed
* MRI, CT or PET-CT of the retroperitoneal space and abdomen at diagnosis is performed
* MRI with the applicator in place at the time of (first) BT will be performed
* Para-aortic metastatic nodes below L1-L2 are allowed
* Patient informed consent

Exclusion Criteria:

* Other primary malignancies except carcinoma in situ of the cervix and basal cell carcinoma of the skin
* Small cell neuroendocrine cancer, melanoma and other rare cancers in the cervix
* Metastatic disease above and beyond the retroperitoneal para-aortic L1-L2 interspace
* Previous pelvic or abdominal radiotherapy
* Previous total or partial hysterectomy
* Combination of preoperative radiotherapy with surgery
* Patients receiving BT only
* Patients receiving EBRT only
* Patients receiving neo-adjuvant chemotherapy or other forms of antineoplastic treatment apart from weekly concomitant cisplatin (40 mg/2). However, adjuvant chemotherapy in the form of 4 courses of 3 weekly Carboplatin (AUC 5) and Paclitaxel (155 mg/m2) is allowed according to departmental policy.
* Contra indications to MRI
* Contra indications to BT

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
local control | 5 years
nodal control | 5 years
systemic control | 5 years
overall survival | 5 years
overall morbidity | 5 years
health-related quality of life: physical functioning | 5 years
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire. Scores ranging from 0 to 100, higher scores indicating better functioning.
health-related quality of life: role functioning | 5 years
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire. Scores ranging from 0 to 100, higher scores indicating better functioning.
health-related quality of life: social functioning | 5 years
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire. Scores ranging from 0 to 100, higher scores indicating better functioning.

SECONDARY OUTCOMES:
cancer specific survival | 5 years
disease specific survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pötter, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official homepage of the EMBRACE study group — https://www.embracestudy.dk/